CLINICAL TRIAL: NCT02338336
Title: A Phase I/II, Two- Staged Randomized, Double-blind Study to Evaluate the Safety and Efficacy of Nowarta110 in Patients With Plantar Warts and Clinical Recovery Successfully Completed
Brief Title: A Phase I/II Double-blind Safety and Efficacy Evaluation of Nowarta110 in Patients With Plantar Warts
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nowarta Biopharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nowarta111545
Record Dates: First submitted 2015-01-10; First posted 2015-01-14 (Estimated); Results first posted 2016-07-19 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-10

CONDITIONS: Plantar Warts

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Nowarta110 3 drops (Experimental): Nowarta110 3 drops administration
  Interventions: Drug: Nowarta110
- Nowarta110 6 drops (Experimental): Nowarta110 6 drops administration
  Interventions: Drug: Nowarta110
- Nowarta110 10 drops (Experimental): Nowarta110 10 drops administration
  Interventions: Drug: Nowarta110

INTERVENTIONS:
Drug: Nowarta110 — Nowarta110 contains fig extract as the main drug substance, and colloidal silver is used as a medium for penetration of fig extract into the wart lesion. Liquid for topical administration.
  Arms: Nowarta110 10 drops; Nowarta110 3 drops; Nowarta110 6 drops
Drug: Placebo — Matching placebo liquid for topic administration.
  Other Names: matching placbo
  Arms: Placebo

SUMMARY:
To evaluate drug safety and efficacy in patients treated with Nowarta110 and to determine therapeutic activity against Plantar Warts

* Clinical Tolerance
* Clinical Recovery
* Evaluate Safety

DETAILED DESCRIPTION:
Plantar Warts occur on the soles (plantar surface of feet) and can be severely debilitating for patients even for normal walking. The severity and magnitude of the warts can vary, but they are the cause of much pain and discomfort for all age groups. Nowarta 110 has been evaluated for the therapy of plantar warts caused by the HPV virus, (HPV infection). Clinical experience in a totals of 124 patients receiving Nowarta 110 for 5 weeks treatment in multiple clinics overseas has demonstrated the potential of Nowarta110 with absolutely no side effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory or recurrent Plantar Warts.
* No wart treatment for the last 12 weeks
* Healthy male or non-pregnant, non-lactating female aged ≥ 18 years or greater
* If female of childbearing potential, use an acceptable form of birth control during the study
* Provide written informed consent or (HIPAA consent/authorization, as applicable

Exclusion Criteria:

* Concurrent medical disorder or disease making implementation or interpretation of the protocol or results difficult or unsafe
* Female subjects who are breast-feeding or planning to become pregnant
* Patients with a history of allergy to silver or fruits
* Subjects with clinically significant unstable medical disorder, life threatening disease, or current malignancies
* Subjects with History of Alcohol abuse or other drug abuse within 2 years prior to Randomization
* Subjects who have been treated with an investigational drug or investigational device within a period of 30 days prior to study enrollment
* Concomitant Medications: any other wart therapy is prohibited during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Iraj E Kiani, Study Chair — Chairman
Locations (1):
- Nowarta Biopharma Inc, Huntington Beach, California, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited at a single center
Pre-assignment Details: Random assignment was stratified by the size of the plantar wart:
  If the lesion size was less than 1 cm2, 3 drops were applied once weekly for 5 weeks If the lesion size was between 1 cm2 and 2 cm2, 6 drops were applied once weekly for 5 weeks If the lesion size was larger than 2 cm2, 10 drops were applied once weekly for 5 weeks
Groups:
- Placebo: Matching Placebo
- Norwarta110 3 Drops: Nowarta110 3 drops administered topically
- Nowarta110 6 Drops: Nowarta110 6 drops administered topically
- Nowarta110 10 Drops: Nowarta110 10 drops administered topically
Period: Overall Study
Arm/Group | Placebo | Norwarta110 3 Drops | Nowarta110 6 Drops | Nowarta110 10 Drops
Started | 26 | 17 | 7 | 4
Completed | 24 | 17 | 7 | 4
Not Completed | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nowarta110: All combined Nowarta110 doses
- Total: Total of all reporting groups
Arm/Group | Placebo | Nowarta110 | Total
Number analyzed (Participants) | 26 | 28 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (10.58) | 34.5 (12.65) | 34.3 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 14 | 11 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 18 | 22 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Lesion Assessment
Description: Lesion (plantar wart) size measured in millimeters. Measurement of the longest dimension was recorded. Observed data
Time Frame: 6 weeks
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- TREATMENT: Nowarta110
Arm/Group | Placebo | TREATMENT
Number analyzed (Participants) | 26 | 28
millimeters
  Baseline | 8.42 (7.229) | 9.14 (6.072)
  Week 1 | 8.42 (7.229) | 8.71 (5.843)
  Week 2 | 7.92 (7.227) | 7.36 (5.864)
  Week 3 | 7.85 (7.182) | 6.00 (4.974)
  Week 4 | 7.58 (7.300) | 4.86 (4.411)
  Week 5 | 7.38 (7.149) | 3.61 (4.076)
  Week 6 | 7.13 (7.267) | 2.25 (4.334)
Statistical Analysis 1: Comparison: Placebo vs TREATMENT; Test type: Superiority or Other; p < 0.001, ANOVA

2. Primary Outcome: Incidence of Zero Lesion Measurement
Description: Percent of participants with lesion measurement either equal to 0 or greater than 0
Time Frame: 6 weeks
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TREATMENT
Number analyzed (Participants) | 26 | 28
percentage of participants
  Lesion Measurement = 0 | 7.7 | 64.3
  Lesion Measurment > 0 | 84.6 | 35.7

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Placebo | Nowarta110
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/28
Other Adverse Events (participants affected / at risk) | 9/26 | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | Nowarta110 (N=28)
Burning/stinging (Skin and subcutaneous tissue disorders) | 9 (9) | 0 (0)
Dryness (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) — Pain on treated area

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No